CLINICAL TRIAL: NCT03629912
Title: Bingocize: A Novel Mobile Application to Help Maintain or Improve Older Adults' Health, Function, and Cognition
Brief Title: Bingocize: A Novel Mobile Application for Older Adult Health
Acronym: Bingocize
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Kentucky University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Matthew Clinton Shake, Associate Professor of Psychological Sciences, Western Kentucky University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 18-048; R15AG055906 (NIH)
Record Dates: First submitted 2018-08-06; First posted 2018-08-14 (Actual); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Activities of Daily Living; Accidental Fall; Sarcopenia; Arteriosclerosis; Diabetes Mellitus, Type 2; Hypertension; Cognitive Decline; Executive Function; Cognitive Aging
MeSH Terms: conditions — Sarcopenia; Arteriosclerosis; Diabetes Mellitus, Type 2; Hypertension; Cognitive Dysfunction | interventions — Aging

STUDY DESIGN:
Intervention Model Description: In each wave of the study (14 weeks per wave), participant groups are randomly assigned to one of four conditions (A,B,C,D). Condition A receives exercise + health education. Condition B receives exercise only. Condition C receives health education only. Condition D receives nothing.
Masking Description: Staff collecting pre- and post-intervention data are masked to participant condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise + Health Education + Bingo (Experimental): Socially-Based Exercise Intervention for Older Adults. Participants use the Bingocize app incorporating exercises AND health information on fall risks + diet/nutrition.
  Interventions: Behavioral: Socially-Based Exercise Intervention for Older Adults
- Exercise + Bingo (Active Comparator): Socially-Based Exercise Intervention for Older Adults. Participants use the Bingocize app incorporating exercises ONLY.
  Interventions: Behavioral: Socially-Based Exercise Intervention for Older Adults
- Health Education + Bingo (Active Comparator): Socially-Based Exercise Intervention for Older Adults. Participants use the Bingocize app incorporating health information on fall risks + diet/nutrition ONLY.
  Interventions: Behavioral: Socially-Based Exercise Intervention for Older Adults
- Bingo Only (No Intervention): Participants use the Bingocize app to play bingo only.

INTERVENTIONS:
Behavioral: Socially-Based Exercise Intervention for Older Adults — A socially-based app that incorporates exercise and/or health education into a format familiar and engaging to older adults, designed to improve adherence to health-promoting behaviors
  Other Names: Bingocize
  Arms: Exercise + Bingo; Exercise + Health Education + Bingo; Health Education + Bingo

SUMMARY:
This study tests the effectiveness of using a new mobile application (Bingocize®) to improve older adults' (a) adherence to an engaging exercise program, and (b) aspects of functional performance, health knowledge, dietary habits, and cognition.

DETAILED DESCRIPTION:
Health-promoting interventions designed to improve physical and mental fitness can help reduce health care costs; they can also help maintain, or even improve, older adults' quality of life. However, getting older adults to adhere to health-promoting exercise interventions remains difficult because such programs are often perceived as being time-consuming, painful, or unenjoyable. The present study's objective is to investigate the effectiveness of a novel technological exercise intervention program for older adults (Bingocize); in doing so, the program has the potential to improve older adults' independence and quality of life. Older adults will participate in a pre/post-intervention design with random assignment to either the experimental or one of three comparison/control groups; each group will play Bingocize in a social setting with other older adults. Participants in the experimental group will use the app to engage in twice-weekly Bingocize sessions for twelve weeks (i.e., Bingo+Exercise+Health Education); control groups will also use the app for twelve weeks but for either health education-only, exercise-only, or bingo-only.

ELIGIBILITY:
Inclusion Criteria:

* Normal or corrected normal vision
* Mobility (i.e., not wheelchair bound)
* English is native language
* Minimum physical standards (e.g., ability to walk at least 10 meters)
* No structured physical activity programs >150 minutes/week in last 6 months

Exclusion Criteria:

* Severe neurological impairments (e.g., Parkinson's)
* Colorblindness
* Dementia

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2022-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew C Shake, PhD, Principal Investigator — Western Kentucky University and Center for Applied Science in Health and Aging; Jason Crandall, PhD, Principal Investigator — Western Kentucky University and Center for Applied Science in Health and Aging
Locations (4):
- United States (4):
  - Webster County Senior Center, Dixon, Kentucky
  - Chester County Senior Center, Henderson, Tennessee
  - Johnson County Senior Center, Johnson City, Tennessee
  - Scotts Hill Senior Center, Scotts Hill, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Time Frame: Data will be available within 6 months after publication, and will remain available for a period of at least 3 years following completion of the clinical trial.
Access Criteria: Investigators whose proposed use of the data has been approved by the Principal Investigators of the clinical trial.
URL: http://www.wku.edu/casha

REFERENCES:
- [Result] Kramer JH, Mungas D, Possin KL, Rankin KP, Boxer AL, Rosen HJ, Bostrom A, Sinha L, Berhel A, Widmeyer M. NIH EXAMINER: conceptualization and development of an executive function battery. J Int Neuropsychol Soc. 2014 Jan;20(1):11-9. doi: 10.1017/S1355617713001094. Epub 2013 Oct 8. PMID 24103232
- [Result] Tinetti ME, Richman D, Powell L. Falls efficacy as a measure of fear of falling. J Gerontol. 1990 Nov;45(6):P239-43. doi: 10.1093/geronj/45.6.p239. PMID 2229948
- See also: Link to Center for Applied Science in Health & Aging — http://www.wku.edu/casha

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twelve participants expressed interest but were then excluded prior to assignment to an arm or group due to failing to meet inclusion criteria.
  Ten participants expressed interest but then prior to assignment to an arm or group, elected to withdraw.
Units Other Than Participants: Senior Center Facility
Groups:
- Exercise + Health Education + Bingo: Socially-Based Exercise Intervention for Older Adults. Participants use the Bingocize app incorporating exercises AND health information on fall risks + diet/nutrition.
  Socially-Based Exercise Intervention for Older Adults: A socially-based app that incorporates exercise and health education into a format familiar and engaging to older adults, designed to improve adherence to health-promoting behaviors
- Exercise + Bingo: Socially-Based Exercise Intervention for Older Adults. Participants use the Bingocize app incorporating exercises ONLY.
  Socially-Based Exercise Intervention for Older Adults: A socially-based app that incorporates exercise into a format familiar and engaging to older adults, designed to improve adherence to health-promoting behaviors
- Health Education + Bingo: Socially-Based Exercise Intervention for Older Adults. Participants use the Bingocize app incorporating health information on fall risks + diet/nutrition ONLY.
  Socially-Based Exercise Intervention for Older Adults: A socially-based app that incorporates health education into a format familiar and engaging to older adults, designed to improve adherence to health-promoting behaviors
Period: Overall Study
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Started | 73; 7 Senior Center Facility | 53; 5 Senior Center Facility | 50; 4 Senior Center Facility | 43; 4 Senior Center Facility
Completed | 44; 7 Senior Center Facility | 40; 5 Senior Center Facility | 41; 4 Senior Center Facility | 39; 4 Senior Center Facility
Not Completed | 29; 0 Senior Center Facility | 13; 0 Senior Center Facility | 9; 0 Senior Center Facility | 4; 0 Senior Center Facility
Not completed — Lost to Follow-up | 19 | 7 | 5 | 1
Not completed — Withdrawal by Subject | 6 | 0 | 1 | 2
Not completed — Illness or Injury Unrelated to Research Study | 3 | 6 | 3 | 1
Not completed — Death | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants with baseline data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only | Total
Number analyzed (Participants) | 73 | 53 | 50 | 43 | 219
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.47 (7.28) | 71.84 (7.71) | 75.04 (6.64) | 70.18 (7.21) | 72.46 (7.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 48 | 39 | 42 | 192
  Male | 10 | 5 | 11 | 1 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 0 | 3
  Not Hispanic or Latino | 63 | 49 | 39 | 40 | 191
  Unknown or Not Reported | 8 | 3 | 11 | 3 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 16 | 0 | 11 | 46
  White | 53 | 33 | 49 | 32 | 167
  More than one race | 0 | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 73 | 53 | 50 | 43 | 219

OUTCOME MEASURES:

1. Primary Outcome: Executive Function Inhibition Measure 1: Flanker Task
Description: Flanker Task designed to measure inhibition, part of the EXAMINER Battery (for scoring method, see References section). EXAMINER generates a score that combines reaction time and accuracy data from the incongruent trials. This scoring method generates accuracy and reaction time sub-scales that range in value between 0 and 5, and the ultimate composite score ranges in value between 0 and 10.
  Minimum=0, Maximum=10, higher = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
score on a scale
  Baseline | 7.30 (1.41) | 7.39 (0.95) | 7.38 (1.18) | 7.51 (1.21)
  Post-Intervention | 7.66 (.80) | 7.54 (.78) | 7.63 (.79) | 7.86 (.62)

2. Primary Outcome: Executive Function Measure: Updating Verbal Working Memory
Description: Dot Counting Task designed to measure verbal working memory, part of the EXAMINER Battery (for scoring method, see References). EXAMINER generates a score is the total number of items correctly recalled across all six trials.
  Minimum=0, Maximum=27, higher = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 43 | 40 | 40 | 39
units on a scale
  Baseline | 21.60 (2.83) | 22.42 (2.43) | 22.50 (2.00) | 21.69 (2.36)
  Post Intervention | 22.56 (2.28) | 22.87 (2.13) | 22.15 (3.10) | 22.12 (2.44)

3. Primary Outcome: Executive Function Measure: Set Shifting Task
Description: Set Shifting Task designed to measure attention during task switching, part of the EXAMINER Battery (for scoring method, see References). EXAMINER generates a score that combines reaction time and accuracy data from the incongruent trials. This scoring method generates accuracy and reaction time sub-scales that range in value between 0 and 5, and the ultimate composite score ranges in value between 0 and 10.
  Minimum=0, Maximum=10, higher = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 40 | 38 | 41 | 37
score on a scale
  Baseline | 6.70 (.93) | 6.51 (1.03) | 6.67 (.94) | 7.05 (.94)
  Post-Intervention | 6.86 (1.07) | 6.82 (.94) | 7.04 (.98) | 7.08 (1.09)

4. Primary Outcome: Executive Function Measure: Verbal Fluency
Description: Verbal Fluency Task designed to measure fluency, part of the EXAMINER Battery (for scoring method, see References). EXAMINER generates a score that represents the total number of words correctly recalled in two tasks: phonemic (letter) and semantic (category).
  Minimum=0, Maximum=unlimited, higher = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
number correct
  Baseline Phonemic Fluency | 9.5 (4.18) | 10.9 (4.39) | 9.04 (3.86) | 10.51 (4.10)
  Post Intervention Phonemic Fluency | 10.34 (5.02) | 9.97 (3.66) | 9.04 (3.91) | 9.25 (3.71)
  Baseline Category Fluency | 10.97 (4.03) | 11.32 (3.35) | 10.73 (3.02) | 11.28 (2.88)
  Post Intervention Category Fluency | 11.06 (3.70) | 11.62 (3.74) | 9.90 (3.24) | 10.97 (2.85)

5. Primary Outcome: Chair Stands: Change in Lower-body Muscular Strength
Description: number of completed chair stands in 30 seconds, minimum=0, higher = better
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: chair stands completed
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 40 | 38 | 39 | 37
chair stands completed
  Baseline | 10.07 (5.24) | 9.28 (4.02) | 9.92 (2.30) | 9.94 (2.26)
  Post Intervention | 11.18 (4.89) | 11.89 (4.11) | 10.87 (3.55) | 10.52 (2.66)

6. Primary Outcome: Change in Dynamic Balance: 360 Degree Turns
Description: 360 degree turns: time to complete. No minimum or maximum value set. Lower = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
seconds
  Baseline | 4.62 (2.88) | 4.07 (1.44) | 3.43 (1.15) | 3.37 (.95)
  Post-Intervention | 4.11 (2.04) | 3.67 (1.57) | 3.53 (1.35) | 3.52 (1.13)

7. Primary Outcome: Executive Function Measure of Inhibition: Continuous Performance Test
Description: Continuance Performance Task is classic response inhibition task, part of the EXAMINER Battery (for scoring method, see References). The score here represents the number of trials out of 100 that the participant responded correctly (i.e., either successfully responded or successfully inhibited a response).
  Minimum=0 Maximum=100, higher = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 43 | 40 | 41 | 39
number correct
  Baseline | 96.76 (5.14) | 96.66 (4.53) | 97.26 (4.94) | 98.17 (2.02)
  Post Intervention | 96.30 (6.35) | 97.92 (2.69) | 97.60 (4.38) | 98.43 (1.65)

8. Secondary Outcome: Crystallized Knowledge of Fall Risks and Proper Diet/Nutrition
Description: Multiple-choice questions constructed by project investigators that cover: recognition of health terms, weight management, proper diet, bone health, environmental fall risks, careful movement. Unit of measure = number correct. Minimum = 0, Maximum = 30. Higher = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
number correct
  Baseline | 19.45 (3.93) | 19.60 (3.96) | 20.07 (3.93) | 20.12 (2.85)
  Post-Intervention | 23.13 (4.30) | 21.67 (3.67) | 23.26 (4.12) | 20.41 (3.46)

9. Secondary Outcome: Grip Strength: Changes in Upper Body Muscular Strength
Description: Grip strength tests using a hand-held dynamometer. No minimum or maximum set. Higher = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
kilograms
  Baseline | 23.34 (7.34) | 24.15 (8.79) | 24.00 (9.60) | 23.56 (6.34)
  Post Intervention | 24.45 (8.98) | 24.80 (7.42) | 24.73 (9.15) | 24.10 (6.17)

10. Secondary Outcome: Fall Efficacy Scale
Description: Self-reported scale assessing confidence in doing activities that may be perceived as having risk for falling (see References).
  Minimum = 10, Maximum = 100. Lower = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
score on a scale
  Baseline | 16.61 (13.12) | 21.00 (20.39) | 19.58 (21.63) | 15.13 (14.22)
  Post Intervention | 17.68 (18.48) | 20.32 (23.46) | 15.65 (16.42) | 15.12 (15.69)

11. Secondary Outcome: Changes in Dietary Habits: Total Added Sugar Intake
Description: Dietary Screener Questionnaire (DSQ) assessing total added sugar intake over past 30 days
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: tsp equivalents
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
tsp equivalents
  Baseline | 13.46 (2.72) | 14.07 (5.30) | 14.94 (6.06) | 14.09 (3.62)
  Post Intervention | 13.28 (4.53) | 13.32 (3.89) | 14.46 (5.10) | 13.79 (3.02)

12. Secondary Outcome: Changes in Quality of Life
Description: CDC Health related quality of life measure item 1 (general health). 1 = Excellent, 5 = Poor. Lower = Better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
units on a scale
  Baseline | 2.95 (.86) | 2.83 (.74) | 2.80 (.92) | 3.00 (.72)
  Post-Intervention | 2.86 (.82) | 2.93 (.79) | 2.83 (.84) | 3.0 (.76)

13. Secondary Outcome: Changes in Weight
Description: Weight calculated by scale measurement
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 43 | 40 | 41 | 39
kg
  Baseline | 84.19 (22.83) | 87.91 (26.60) | 78.11 (14.45) | 86.79 (21.82)
  Post Intervention | 84.09 (22.11) | 86.83 (22.67) | 80.00 (15.93) | 86.27 (21.37)

14. Secondary Outcome: Systolic Blood Pressure
Description: Systolic Blood pressure calculated by sphygmomanometer.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
mmHg
  Baseline | 135.23 (12.99) | 134.03 (13.97) | 136.12 (13.64) | 135.18 (12.42)
  Post Intervention | 136.25 (16.63) | 143.21 (10.71) | 141.83 (19.02) | 141.21 (22.10)

15. Secondary Outcome: Diastolic Blood Pressure
Description: Diastolic Blood pressure calculated by sphygmomanometer
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
mmHg
  Baseline | 75.07 (10.04) | 78.23 (8.87) | 76.12 (7.68) | 75.54 (7.33)
  Post Intervention | 77.14 (9.17) | 79.61 (11.03) | 77.83 (10.39) | 79.85 (9.07)

16. Primary Outcome: Timed Up and Go (TUG) Test: Change in Dynamic Balance
Description: Timed Up and Go (TUG) Test used to assess mobility and risk for falling. Number of seconds needed to stand up from a chair, walk 10 feet, turn around, walk back 10 feet, and sit back down in chair. No minimum or maximum value is set. Lower = better.
Time Frame: Baseline and 12 Weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
Number analyzed (Participants) | 44 | 40 | 41 | 39
seconds
  Baseline | 12.58 (6.57) | 12.51 (4.49) | 11.12 (2.72) | 10.96 (2.98)
  Post-Intervention | 12.44 (6.48) | 11.78 (4.72) | 10.49 (3.13) | 11.57 (2.96)

ADVERSE EVENTS:
Time Frame: Twice weekly during 1 hour program sessions, for a duration of 12 weeks
Arm/Group | Exercise + Health Education + Bingo | Exercise + Bingo | Health Education + Bingo | Bingo Only
All-Cause Mortality (participants affected / at risk) | 1/73 | 0/53 | 0/50 | 0/43
Serious Adverse Events (participants affected / at risk) | 3/73 | 6/53 | 3/50 | 1/43
Other Adverse Events (participants affected / at risk) | 0/73 | 0/53 | 0/50 | 0/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Exercise + Health Education + Bingo (N=73) | Exercise + Bingo (N=53) | Health Education + Bingo (N=50) | Bingo Only (N=43)
Cancer Diagnosis (General disorders) | 0 | 0 | 0 | 1
Aneuryism (Vascular disorders) | 0 | 0 | 1 | 0
Wrist Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Edema (Vascular disorders) | 0 | 1 | 0 | 0
Unspecified Health Issues (General disorders) | 2 | 4 | 2 | 0
stroke (Vascular disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
COVID-19 Pandemic began in the Middle of this Intervention, resulting in the loss of approximately 35-40% of the overall participant sample who were in the middle of the clinical trial intervention and had to withdraw from the study. Other data collection waves were started and completed before the pandemic, or started and completed after the pandemic, which introduces the possibility of history effects impacting interpretations of the data from participants who did complete the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03629912/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/12/NCT03629912/ICF_001.pdf